CLINICAL TRIAL: NCT00934492
Title: Randomized, Placebo Controlled Trial of Cotrimoxazole Prophylaxis Amongst HIV-uninfected Children With Severe Malnutrition
Brief Title: Cotrimoxazole Prophylaxis in Severely Malnourished Children
Acronym: CTX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SSC 1562; OXTREC 18 09; WT 083579
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Nutrition Disorders; Life-threatening Infection
Keywords: Malnutrition; Wasting; Kwashiorkor; Immune deficiency; Infection; Prophylaxis; Mortality; Kenya
MeSH Terms: conditions — Nutrition Disorders; Malnutrition; Cachexia; Kwashiorkor; Immunologic Deficiency Syndromes; Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cotrimoxazole dispersible tablet (Active Comparator): Children between 2-6 months will receive single dispersible tablet of 120mg,daily while children over 6 months to 5 years will receive 240 mg dispersible tablet daily for six months.
  Interventions: Drug: Cotrimoxazole dispersible tablet
- Placebo dispersible tablet (Placebo Comparator): Children between 2-6 months will receive single dispersible Placebo tablet of 120mg,daily while children over 6 months to 5 years will receive 240 mg dispersible Placebo tablet daily for six months.
  Interventions: Drug: Placebo dispersible tablet

INTERVENTIONS:
Drug: Cotrimoxazole dispersible tablet — Cotrimoxazole dispersible tablets 120/240mg daily for six consecutive months.
  Other Names: Cosatrim; Septrin; Bactrim
  Arms: Cotrimoxazole dispersible tablet
Drug: Placebo dispersible tablet — Placebo dispersible tablets 120/240mg daily for six consecutive months.
  Other Names: Placebo
  Arms: Placebo dispersible tablet

SUMMARY:
This trial aims to test the hypothesis that mortality among Kenyan children with severe malnutrition following initial stabilisation is due to ongoing vulnerability to infectious disease, and that long term daily co-trimoxazole prophylaxis will reduce mortality.

The objective is to conduct a randomized, double blind, placebo-controlled trial of cotrimoxazole prophylaxis for 6 months among HIV-uninfected children with severe malnutrition following stabilization. The primary outcome will be survival at one year. Secondary outcomes are toxicity, growth, the frequency and causes of hospitalisation and microbial resistance to antibiotics.

Cotrimoxazole has striking protective efficacy against mortality among children with HIV, despite not altering the underlying immune deficiency. It is hypothesised that co-trimoxazole prophylaxis will have a similar effect in children immunocompromised because of severe malnutrition. Worldwide, severe malnutrition is commoner than HIV in childhood and co-trimoxazole is cheap and widely available, making it easily translatable to policy.

DETAILED DESCRIPTION:
Malnutrition is the most important underlying risk factor for childhood death in developing countries. Severely malnourished children are at greatly increased risk of death from infectious diseases in the community, in hospital and following discharge. Malnutrition and infection are synergistic, in part because malnutrition causes secondary immune deficiency, whilst infections cause losses and diversion of nutrients. This synergy is exacerbated by a high level of exposure to pathogens. Among children treated for severe malnutrition in Africa, mortality following discharge from hospitals ranges between 8% and 41%.

Cotrimoxazole is a synthetic antibacterial combination that blocks two steps of folate metabolism involved in the biosynthesis of nucleic acids and proteins essential to many bacteria and some parasites, including Plasmodium falciparum. It is cheap, widely available and has an established safety profile in African populations. Cotrimoxazole prophylaxis dramatically reduces mortality among children with HIV, irrespective of the degree of immune suppression. The primary effect is in reducing bacterial infection, especially pneumonia. the effect has been demonstrated in areas with high levels of cotrimoxazole resistance bacteria. It is also widely used in developed countries among children with other immune deficiencies to prevent infection. Children with severe malnutrition are immune deficient, as evidenced by their susceptibility to infectious diseases, and may therefore benefit from daily antimicrobial prophylaxis.

The objective is to conduct a randomized, double blind, placebo-controlled trial of cotrimoxazole prophylaxis for 6 months among HIV-uninfected children with severe malnutrition following stabilization. The primary outcome will be survival at one year. Secondary outcomes are toxicity, growth, hospitalisation, microbial resistance in carriage and pathogenic organisms and markers of inflammation and immune function.

On 26th September 2012, on advice from an independent senior statistician who reviewed the actual event rate in the control arm, the rates of recruitment and loss to follow up, the Trial Steering Committee recommended that the trial team to recruit at least 1750 participants to achieve the original objective of having >90% power to detect a reduction in mortality during 12 months follow up of 33%. Recruitment was stopped on 31st March 2013 at 1781 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 months to 5 years
* Admitted to hospital
* Severe malnutrition: age 6 months to 5 years: MUAC <11cm; age 2 to 6 months: MUAC for age <-3 z scores compared to the WHO growth standards; or kwashiorkor at any age (defined in current WHO guidelines) for enrollments up to 24th March 2011.
* Severe malnutrition:age 6 months to 5 years: MUAC <11.5cm; age 2 to 6 months: MUAC <11.0cm; or kwashiorkor at any age (defined in current WHO guidelines) for enrollments from 24th March 2011, following protocol amendment.
* HIV rapid test negative, or if under 18 months, PCR negative and no longer breastfeeding for at least 6 weeks
* Planning to remain within study area and willing to come for all protocol specified visits

Exclusion Criteria:

* Refusal to give informed consent
* Cotrimoxazole is specifically contra-indicated (e.g. porphyria)
* Known hypersensitivity reaction to sulpha drugs or trimethoprim

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1781 (Actual)
Dates: Start 2009-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Mortality | 12 months

SECONDARY OUTCOMES:
Frequency and causes of hospital re-admission | 12 months
Growth | 12 months
Microbial population and antimicrobial resistance | 12 months
Immune activation and inflammatory markers; markers of immune function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James A Berkley, FRCPCH, Principal Investigator — Universitiy of Oxford & Kenya Medical Research Institute
Locations (4):
- Kenya (4):
  - KEMRI/Wellcome Trust Research Programme, Kilifi, Coast
  - Malindi District Hospital, Malindi, Coast
  - Coast Provincial General Hospital, Mombasa, Coast
  - Mbagathi District Hospital, Nairobi

REFERENCES:
- [Derived] Ngari MM, Iversen PO, Thitiri J, Mwalekwa L, Timbwa M, Fegan GW, Berkley JA. Linear growth following complicated severe malnutrition: 1-year follow-up cohort of Kenyan children. Arch Dis Child. 2019 Mar;104(3):229-235. doi: 10.1136/archdischild-2018-315641. Epub 2018 Sep 28. PMID 30266874
- [Derived] Ngari MM, Mwalekwa L, Timbwa M, Hamid F, Ali R, Iversen PO, Fegan GW, Berkley JA. Changes in susceptibility to life-threatening infections after treatment for complicated severe malnutrition in Kenya. Am J Clin Nutr. 2018 Apr 1;107(4):626-634. doi: 10.1093/ajcn/nqy007. PMID 29635501
- [Derived] Ngari MM, Thitiri J, Mwalekwa L, Timbwa M, Iversen PO, Fegan GW, Berkley JA. The impact of rickets on growth and morbidity during recovery among children with complicated severe acute malnutrition in Kenya: A cohort study. Matern Child Nutr. 2018 Apr;14(2):e12569. doi: 10.1111/mcn.12569. Epub 2017 Nov 27. PMID 29178404
- [Derived] Berkley JA, Ngari M, Thitiri J, Mwalekwa L, Timbwa M, Hamid F, Ali R, Shangala J, Mturi N, Jones KD, Alphan H, Mutai B, Bandika V, Hemed T, Awuondo K, Morpeth S, Kariuki S, Fegan G. Daily co-trimoxazole prophylaxis to prevent mortality in children with complicated severe acute malnutrition: a multicentre, double-blind, randomised placebo-controlled trial. Lancet Glob Health. 2016 Jul;4(7):e464-73. doi: 10.1016/S2214-109X(16)30096-1. Epub 2016 Jun 2. PMID 27265353